CLINICAL TRIAL: NCT02421029
Title: Prolonged Gadolinium Retention After MRI Imaging in Patients With Normal Renal Function
Brief Title: Prolonged Gadolinium Retention After MRI Imaging
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: it was logistically difficult to obtain the drug needed to conduct the study
Sponsor: Mt. Sinai Medical Center, Miami (Other)
Responsible Party: Principal Investigator, Gervasio Lamas, MD, Chair, Department of Medicine, Mt. Sinai Medical Center, Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MRI-EDTA
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Heavy Metal Toxicity
Keywords: gadolinium; calcium disodium ethylenediaminetetraacetic acid (EDTA); heavy metal toxicity
MeSH Terms: conditions — Heavy Metal Poisoning | interventions — Pentetic Acid; Edetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- edetate calcium disodium (Experimental): Subjects who had a gadolinium-enhanced MRI within 1-4 weeks or within 3-6 months before enrollment will receive a single dose of edetate calcium disodium to evaluate levels of gadolinium in their urine, pre and post infusion.
  Interventions: Drug: edetate calcium disodium

INTERVENTIONS:
Drug: edetate calcium disodium — All subjects will receive a 250 mL 5% dextrose intravenous infusion over 1 hour that contains 1 gr of edetate calcium disodium
  Other Names: Calcium Disodium Versenate

SUMMARY:
The researchers propose to investigate the prevalence of gadolinium in the urine of patients with a prior gadolinium-enhanced MRI before and after a edetate calcium disodium challenge. Moreover, will investigate if there is any correlation of gadolinium urine levels with levels of endogenous (e.g zinc) and xenobiotic metals.

DETAILED DESCRIPTION:
The investigators propose to enroll 20 volunteers in this pilot study, including males older than 20 years and postmenopausal women in two groups: Group 1: Individuals who had a gadolinium-enhanced MRI study within 1-4 weeks before participation and Group 2: Individuals who had gadolinium-enhanced MRI study within 3-6 months before enrollment. The results will inform future analyses of gadolinium retention, excretion, and potential symptoms associated with same.

Thus, the specific aims of this cross sectional study are to:

1. Evaluate levels of gadolinium in the urine of adults with normal kidney function and a prior MRI performed within 6 months at baseline, and after a single dose of edetate calcium disodium .
2. Evaluate levels of endogenous and xenobiotic metal levels and their relationship with gadolinium levels.
3. Evaluate for symptoms of gadolinium toxicity.

ELIGIBILITY:
Inclusion Criteria:

• Subjects who had a contrast enhanced MRI for any indication within 1-4 weeks or 3-6 months, and normal renal function assessed by normal glomerular filtration rate (GFR) >60 mL/min/1.73 m2 at the time of the gadolinium-enhanced MRI study.

Exclusion Criteria:

* Allergy to edetate calcium disodium
* Prior chelation therapy with edetate disodium since the administration of gadolinium
* Blood pressure >160/100
* No venous access
* Platelet count <100,000/mm3
* Liver disease or alanine transaminase (ALT) or aspartate transaminase (AST) >2.0 times the upper limit of normal
* Diseases of copper, iron, or calcium metabolism
* Women of child-bearing potential
* History of lead intoxication; lead encephalopathy; cerebral edema.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
gadolinium levels in urine before and after an edetate calcium disodium challenge | within 6 months of a gadolinium-enhanced MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Medical Center, Miami Beach, Florida, United States